CLINICAL TRIAL: NCT03321292
Title: Effect of L-Arginine on Intrauterine Growth Restriction Fetuses Measured by Birth Weight: Randomized Controlled Trial
Brief Title: L-arginine in Treatment of Intrauterine Growth Restriction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hayam Fathy Mohammad, Assistant Professor of Obstetrics and Gynecology , Ain Shams University, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hayam Fathy Mohammad 2
Record Dates: First submitted 2017-09-28; First posted 2017-10-25 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Intrauterine Growth Restriction Asymmetrical
MeSH Terms: interventions — Arginine; Tablets; Aspirin

STUDY DESIGN:
Intervention Model Description: Group(A) 130 pregnant women diagnosed with IUGR will receive L-arginine and Acetylesalicylic acid 75mg Group(B) 130 pregnant women diagnosed with IUGR will receive Acetylesalicylic acid 75mg
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-arginine and Acetylesalicylic acid (Experimental): L-arginine 1000mg capsules( manufactured by Putriant Pride,INC Holbrook,NY 11741 U.S.A.) every 8 hours Acetylesalicylic acid 75 mg tablet(manufactured by Multi_Apex Pharma , Egypt) once daily will be given for patients of group A starting from diagnosis till birth
  Interventions: Drug: L-arginine 1000 mg and Acetylesalicylic acid75mg
- Acetylesalicylic acid75mg (Active Comparator): acetylsalicylic acid 75 mg tablet(manufactured by Multi_Apex Pharma , Egypt) orally once daily will be given for patients of group B starting from diagnosis till birth
  Interventions: Drug: acetylsalicylic acid 75 mg

INTERVENTIONS:
Drug: L-arginine 1000 mg and Acetylesalicylic acid75mg — l-arginine 1000mg capsule will be given every 8 hours till delivery and acetylesalicylic acid75mg tablet once starting of diagnosis till birth.
  Other Names: L- arginine 1000mg capsule and Ezacard 75 mg tablet
  Arms: L-arginine and Acetylesalicylic acid
Drug: acetylsalicylic acid 75 mg — acetylsalicylic acid 75 mg will be given orally once daily for group B starting of diagnosis till birth.
  Other Names: Ezacard 75mg
  Arms: Acetylesalicylic acid75mg

SUMMARY:
Intrauterine growth restriction is an important problem in neonatal care. Intrauterine growth restriction (IUGR) is defined as a fetal weight below the 10th percentile for gestational age. One of the main causes of IUGR is placental insufficiency.

Nitric oxide(NO) increases placental blood flow. So,it might be useful to improve IUGR pregnancy outcome .

DETAILED DESCRIPTION:
The study population includes pregnant women attending Antenatal care clinic of Ain Shams University Maternity Hospital who first time diagnosed of IUGR at our antenatal care outpatient clinic either referred for this cause After confirm diagnosis of IUGR and distributing patient into two groups Patient in first group will receive oral L-arginine 3000mg/day till delivery and Acetylesalicylic acid 75mg once daily.

Patients in second group will receive Acetylesalicylic acid 75mg once daily. then follow up of both group by:

1. Daily fetal movement counting
2. Day after day CTG
3. Doppler twice weekly
4. Pelvic u/s weekly for:

A) Head circumference, Abdominal circumference, femur length B) Fetal weight C) Liquor amount: Amniotic Fluid Index Or MeanVertical Pocket

Decision of delivery will be determined when:

A) Fetal distress (non stress CTG) B) Mother starts labour C) Reversed umbilical artery Doppler.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women diagnosed with IUGR from 28 weeks
* Singleton pregnancy
* No maternal systemic disease
* No congenital fetal malformation
* Estimated fetal weight below 10th percentile

Exclusion Criteria:

* All pregnant woman diagnosed with IUGR before 28 weeks
* Multiple pregnancy
* Maternal systemic disease
* Congenital fetal malformation

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 260 (Estimated)
Dates: Start 2017-10-15 (Actual); Primary Completion 2018-12-01 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
Birth weight | 15 min
  neonatal birth weight will be measured immediately following delivery and compared with the estimated fetal weight measured by ultrasound

SECONDARY OUTCOMES:
Apgar score | at one and five minute after birth.
  The Apgar scale is determined by evaluating the newborn baby on five simple criteria on a scale from zero to two, then summing up the five values thus obtained. The resulting Apgar score ranges from zero to 10. The five criteria are (Appearance, Pulse, Grimace, Activity, Respiration).
Amniotic fluid index | evey one week from 28 weeks gestation till 40 weeks gestation
  Amniotic fluid index (sum of the vertical diameter of the four pocket of amniotic fluid )
Umbilical artery Doppler | every from 28 weeks gestation till 40 weeks gestation
  umbilical artery Doppler will measured by two dimensional ultrasound power Doppler twice weekly for the presence of any abnormality as: marked decreased diastolic blood flow, absent or reversed diastolic blood flow.

CONTACTS AND LOCATIONS:
Overall Officials: Hayam FA Mohammad, MD, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt